CLINICAL TRIAL: NCT03866252
Title: LSD Therapy for Persons Suffering From Major Depression: A Randomised, Double-blind, Active-placebo Controlled Phase II Study
Brief Title: LSD Therapy for Persons Suffering From Major Depression
Acronym: LAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Department of Psychiatry Basel (UPK Basel; Prof. Dr. med. Stefan Borgwardt) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BASEC 2018-02370
Record Dates: First submitted 2019-02-08; First posted 2019-03-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Subjects in the treatment arm will receive 100 μg LSD (first session) and 100 or 200 μg LSD (second session) per os.
  Interventions: Drug: LSD
- Control Arm (Active Comparator): Subjects in the control arm will receive 25 μg LSD (first session) and 25 μg LSD (second session) per os.
  Interventions: Drug: LSD

INTERVENTIONS:
Drug: LSD — LSD administration per os
  Other Names: Lysergic Acid Diethylamide

SUMMARY:
Background: Major Depressive Disorder is one of the most prevalent mental illnesses, leading to substantial personal distress and economical consequences. Pharmacological Treatment is limited and relapse is frequent.

Lysergic acid diethylamide (LSD) was extensively investigated in humans in the 1950s and 1960s and was shown to attenuate depressive symptoms. Clinical research with LSD ended in the 1970s due to regulatory restrictions but its use for personal and recreational purposes continued. In recent years, there has been a renewed interest in the use of hallucinogens in psychiatric research and practices, reconsidering LSD's antidepressant potential. Larger, well-designed and placebo-controlled studies are warranted. This study will evaluate the potential benefits of LSD-assisted psychotherapy in patients suffering from Major Depressive Disorder.

Objective: To test the efficacy of LSD in patients with Major Depressive Disorder.

Design: Randomised, double-blind, active-placebo-controlled trial using either two moderate to high doses of LSD (100 µg and 100 µg or 100 µg and 200 µg) as intervention and two low doses of LSD (25 µg and 25 µg) as active-placebo control.

Participants: 60 patients aged > 25 years with Major Depressive Disorder (according to DSM-V).

Main outcome measures: Change in depressive symptomatology (IDS, BDI), anxiety (STAI), and general psychopathology (SCL-90) compared with active-placebo-assisted psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* > 25 years
* Sufficient understanding of the German language

Exclusion Criteria:

* < 25 years
* Concomitant diagnosis of past or present psychotic disorder
* Concomitant diagnosis of past or present bipolar disorder
* First degree relative with a psychotic disorder
* Unable or unwilling to discontinue antidepressant medication
* Pregnancy or breastfeeding
* Known hypersensitivity to LSD
* Somatic disorders including central nervous system (CNS) involvement
* Known or suspected non-compliance, drug or alcohol abuse
* Metal implants
* Weight < 42 kg
* Suicide risk or very likely to require psychiatric hospitalisation

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms assessed by questionnaire compared with active placebo | Baseline; 1 week before first intervention; 2 weeks after first intervention; 2, 6, and 12 weeks after LSD
  Inventory of Depressive Symptomatology (IDS-C, clinician-rated). Scores are obtained by summing responses to the items, with a total score ranging from 0 to 84 and higher scores indicating more and/or stronger depressive symptoms.
Change in depressive symptoms assessed by questionnaire compared with active placebo | Baseline; 1 week before first intervention; 2 weeks after first intervention; 2, 6, and 12 weeks after LSD
  Inventory of Depressive Symptomatology (IDS-SR, self-rated). Scores are obtained by summing responses to the items, with a total score ranging from 0 to 84 and higher scores indicating more and/or stronger depressive symptoms.

OTHER OUTCOMES:
Change in depressive symptoms assessed by questionnaire compared with active placebo | Baseline; 1 week before first intervention; 2 weeks after first intervention; 2, 6, and 12 weeks after LSD
  Beck Depression Inventory (BDI). Scores are obtained by summing responses to the items, with a total score ranging from 0 to 63 and higher scores indicating more and/or stronger depressive symptoms.
Changes in state and trait anxiety assessed by questionnaire compared with active placebo | Baseline; 2 weeks post-intervention
  State-Trait Anxiety Inventory (STAI). State and trait anxiety are being assessed separately. Each type of anxiety is being represented by 20 different items. Scores range from 20 to 80, with higher scores indicating greater anxiety.
Changes in general psychopathology assessed by questionnaire compared with active placebo | Baseline; 1 week before first intervention; 2 weeks after first intervention; 2, 6, and 12 weeks after LSD
  Symptom Check List (SCL-90, 90-item version). Consists of 9 subscales investigating psychopathological symptoms (somatization, obsessive-compulsivity, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism), offering five answers (i.e. not at all, a little, fairly, a lot, extremely). SCL-90 total score = 360; subscale total score = 40. Higher scores indicate greater psychological impairment.
Changes in existential anxiety assessed by questionnaire compared with active placebo | Baseline; 2 weeks after first treatment; 2 weeks after second treatment
  Existential Concerns Questionnaire (EAQ). Item scores are assessed in a yes/no format.
Changes in mindfulness assessed by questionnaire compared with active placebo | Baseline; 2 weeks after first treatment; 2 weeks after second treatment
  Five Facet Mindfulness Questionnaire (FFMQ). Item scores are assessed on a scale from 1 (never) to 5 (very often or always). Higher scores indicate higher greater levels of mindfulness.
Changes in humility assessed by questionnaire compared with active placebo | Baseline; 6 weeks post-treatment
  Elliot Humility Scale (EHS). Item scores are assessed on a scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher greater levels of humility.
Changes in humility assessed by questionnaire | Baseline; 6 weeks post-treatment compared with active placebo
  Jankowski Humility Scale (JHS). Item scores are assessed on a scale from 1 (not at all) to 5 (absolutely). Higher scores indicate higher greater levels of humility.
Changes in the personality trait "absorption" assessed by questionnaire compared with active placebo | Baseline
  Tellegen Absorption Scale (TAS). Item scores are assessed on a scale from 0 (not at all) to 4 (absolutely). Higher scores indicate higher greater levels of trait absorption.
Acute subjective effects assessed via questionnaire compared with active placebo | At weeks 3 and 7
  The Visual Analog Scale (VAS). Items assess acute subjective drug effects (e.g. intensity, liking) Item scores are assessed on a visual scale ranging from 1% to 100%. Higher scores indicate greater subjective effects.
Characteristics of altered states of consciousness assessed by questionnaire | At weeks 3 and 7
  States of Consciousness Questionnaire (SCQ). Items retrospectively assess subjective drug effects. Item scores are assessed on a scale ranging from 0 to 5. Higher scores indicate greater subjective effects associated with a different state of consciousness.
Characteristics of altered states of consciousness assessed by questionnaire compared with active placebo | At weeks 3 and 7
  5-Dimensional Altered States of Consciousness Questionnaire (5D-ASC). Items retrospectively assess subjective drug effects. Item scores are assessed on a visual scale ranging from 1% to 100%. Higher scores indicate greater subjective effects associated with a different state of consciousness.
Changes in mystical-type experiences assessed by questionnaire | Baseline; 6 weeks post-treatment compared with active placebo
  Mysticism Scale (MS). Item scores are assessed on a scale ranging from +4 (extremely accurate) to -4 (extremely inappropriate). Higher scores indicate greater levels of mystical experiences.
Acquisition of physical conditions / complaints assessed by questionnaire | Baseline; at weeks 2, 3, 5, 7, 9, 13
  List of complaints (LC). Assesses acute complaints (e.g. pain, coughing, nausea) in a yes/no frmat. A higher number of "yes" answers indicates more complaints. Total "yes" score ranges from 0 to 65.
Perception of therapeutic alliance assessed by questionnaire | 1 week pre-treatment
  Helping Alliance Questionnaire (therapist version (HAQ-T), patient version (HAQ-P). Item scores are assessed on a scale ranging from 1 (very accurate) to 6 (very inaccurate). Lower scores indicate increased subjective helping alliance.
Subjective evaluation of mood assessed by questionnaire | Baseline; at weeks 2, 3, 5, 7, 9, 13
  Adjective Mood Rating Scale (clinician version (AMRS-C), patient version (AMRS-P). Scale consists of 60 adjectives describing different moods (e.g. "nervous", "concentrated", "drowsy"), offering four response possibilities (i.e. not at all, a little, fairly, strongly). Items are analyzed separately.
Assessment of personality by questionnaire | Baseline
  NEO-Five-Factor-Inventory (NEO-FFI). The NEO-FFI assesses five personality traits (i.e. neuroticism, extraversion, openness, agreeableness and conscientiousness) on a scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher manifestation of a particulare personality trait.
Assessment of religiosity by questionnaire | Baseline
  Religiosity Scale (Z-Scale). This 7-item scale assesses the degree of religiosity on ascending scales ranging from "not at all" to "very often". Higher scores indicate higher levels of religiosity.
Persisting effects of treatment assessed by questionnaire | 12 weeks post-treatment
  Persisting Effects Questionnaire (PEQ). Scores are assessed on a scale from 0 (not at all) to 5 (extremely). Higher scores (under consideration of reverse-scored items) indicate stronger persisting treatment effects.
Changes in brain-derived neurotrophic factor (BDNF) | One day and 12 weeks post-treatment
  Changes in brain-derived neurotrophic factor as measured by blood concentrations compared with active placebo
Changes in hypothalamic-pituitary-adrenal (HPA) axis function | 2 weeks post-treatment
  Changes in hypothalamic-pituitary-adrenal (HPA) axis function as measured with salivary cortisol awakening responses compared with active placebo
Changes in immunoregulation and Inflammation compared with active placebo | One day and 12 weeks post-treatment
  Measured via blood levels of macrophage migration inhibitory factor and interleukin-1 beta
Brain activation during fearful face processing and working memory processing compared with placebo | One week pre-treatment and one day post-treatment
  Functional Magnetic Resonance Imaging (fMRI)
Brain Perfusion in treatment condition compared with active placebo | One week pre-treatment and one day post-treatment
  Diffusion Tensor Imaging (DTI)
Brain Perfusion compared with active placebo | One week pre-treatment and one day post-treatment
  Arterial Spin Labeling (ASL)
Changes in sleep patterns | From one week pre-treatment to two weeks post-treatment
  Actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Felix Müller, MD, Study Chair — Department of Psychiatry
Locations (1):
- Universitäre Psychiatrische Kliniken, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Muller F, Zaczek H, Becker AM, Ley L, Borgwardt S, Santos de Jesus J, Loh N, Kohut J, Auernig M, Boehlke C, Liechti ME. Efficacy and safety of low- versus high-dose-LSD-assisted therapy in patients with major depression: A randomized trial. Med. 2025 Sep 12;6(9):100725. doi: 10.1016/j.medj.2025.100725. Epub 2025 Jun 6. PMID 40482648